CLINICAL TRIAL: NCT00073619
Title: Community Violence and Youth: Preventing Anxiety Disorders
Brief Title: Preventing Anxiety Disorders in Urban Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH063143 (NIH); R21MH063143 (NIH); DSIR CT-P (Other: NIMH)
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Anxiety Disorders
Keywords: Violence; School based; Urban Youth; Prevention; Community
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral group therapy (Experimental): School-based anxiety preventive intervention (cognitive-behavioral group therapy) originally designed for Australian children that was culturally and contextually modified for inner-city children exposed to community violence. Participants received the weekly intervention and rewards for participating in the assessments.
  Interventions: Behavioral: Cognitive-behavioral group therapy
- Non-intervention Comparison (No Intervention): Provide no active intervention to the comparison group, although assess the children at the same assessment points as the experimental group. Participants in the control arm were told they were FRIENDS Program participants.They received rewards for participating in the assessments.

INTERVENTIONS:
Behavioral: Cognitive-behavioral group therapy — School-based anxiety preventive intervention (cognitive-behavioral group therapy) originally designed for Australian children that was culturally and contextually modified for inner-city children exposed to community violence. Participants received the weekly intervention and rewards for participating in the assessments.
  Arms: Cognitive-behavioral group therapy

SUMMARY:
This study will determine the effectiveness of a cognitive-behavioral group therapy program in preventing anxiety disorders in at-risk children exposed to community violence.

DETAILED DESCRIPTION:
Community violence is a major public health problem in low-income, urban communities. The mental health impact of living in a violent community is significant, particularly for children. Community violence exposure is associated with various symptoms of anxiety. Unfortunately, little research on the prevention of community-related anxiety in youth has been conducted. This study involves a school-based prevention and cognitive behavioral therapy program that will involve predominantly African American children who live in urban areas and are at risk for developing anxiety disorders.

Children in this study will be randomly assigned to either an anxiety prevention and early intervention group or a nonintervention group for approximately 3 months. Child, parent, and teacher assessments of anxiety symptoms will be made at the end of the study and at a 6-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Mild exposure to community violence
* Mild to moderate anxiety symptoms or disorders
* Attending public elementary school in an urban area
* In 3rd to 5th grades

Exclusion Criteria:

* Diagnostic and Statistical Manual-IV disruptive behavior disorder
* Too many or too few anxiety symptoms

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2001-12; Primary Completion 2007-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Revised Children's Manifest Anxiety Scale | Past month
  Revised Children's Manifest Anxiety Scale (RCMAS; Reynolds & Richmond, 1997), a self-report measure of the level and nature of anxiety in children and adolescents. It is a 37-item questionnaire in which students agree or disagree to statements pertaining to how some people think or feel about themselves, assessing different ways anxiety is manifested. A higher score indicates more anxiety and distress. The RCMAS has good internal consistency (alpha = 0.83) and test-retest reliability (r = 0.68). In the FRIENDS study, Total RCMAS reliability was alpha = 0.83 at baseline and alpha = 0.84 at post-assessment.

SECONDARY OUTCOMES:
Wechsler Individual Achievement Test-Screener | Past year
  Academic achievement was assessed using the Wechsler Individual Achievement Test-Screener (WIAT-Screener; Psychological Corporation, 1992), which consists of three subtests of the comprehensive WIAT battery (i.e., Basic Reading, Mathematics Reasoning, Spelling). It assesses basic academic skills; permits the calculation of age- and grade-based standard scores; was standardized using a large representative sample; is widely used; and has demonstrated reliability and validity with little evidence of practice effects (Psychological Corporation, 1992).
Multicultural Events Schedule for Adolescents | Past year
  Adverse life events were assessed using the Multicultural Events Schedule for Adolescents (MESA; Gonzales, Gunnoe, Samaniego, & Jackson, 1995), developed to assess major and minor life events specific to an urban multiethnic population (Gonzales et al., 1995). It was normed on African American, European American, and English- and Spanish-speaking Mexican Americans. The MESA includes 84 items in which a student responds yes or no to each life events over the past year. A Total life events score is based on the number of events endorsed, with a higher score indicating more adverse life events and hassles. The MESA has adequate concurrent validity and test-retest reliability (Gonzales et al., 1995). In the FRIENDS project, the MESA Total score alpha = .89 at baseline, and alpha = .95 at the post-assessment.
Children's Report of Exposure to Violence | Past year and Lifetime
  Children's Report of Exposure to Violence (CREV; Cooley, Turner, & Beidel, 1995). The CREV is a widely used self-report questionnaire developed to assess children's lifetime exposure to community violence. It has good two-week test-retest reliability (r = 0.75), internal consistency (overall alpha = .78), and construct validity (Cooley et al., 1995). Twenty-nine scored CREV items are rated on a 5-point Likert scale, ranging from 0-''no, never'' to 4-''everyday,'' to indicate the frequency of exposure to community violence via four modes (i.e., media, hearsay, witness, victimization). Types of violent situations include being chased or threatened, beaten up, robbed or mugged, shot, stabbed, or killed. Higher scores indicate more perceived exposure. A past-year version of the CREV was developed and administered at the post-assessment evaluation. Cronbach's alpha for the lifetime CREV Total score was .88 at baseline and .90 for the past-year version.

CONTACTS AND LOCATIONS:
Overall Officials: Michele R Cooley, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Background] Lambert SF, Cooley MR, Campbell KD, Benoit MZ, Stansbury R. Assessing anxiety sensitivity in inner-city African American children: psychometric properties of the childhood anxiety sensitivity index. J Clin Child Adolesc Psychol. 2004 Jun;33(2):248-59. doi: 10.1207/s15374424jccp3302_5. PMID 15136188
- [Background] Cooley MR, Boyce CA. An introduction to assessing anxiety in child and adolescent multiethnic populations: challenges and opportunities for enhancing knowledge and practice. J Clin Child Adolesc Psychol. 2004 Jun;33(2):210-5. doi: 10.1207/s15374424jccp3302_1. PMID 15136184
- [Result] Cooley, M., Boyd, R.C., & Grados, J.J. (2004). Feasibility of an anxiety preventive intervention for community violence exposed children. The Journal of Primary Prevention, 25(1), 105-123.
- [Result] Cooley-Strickland MR, Griffin RS, Darney D, Otte K, Ko J. Urban African American youth exposed to community violence: a school-based anxiety preventive intervention efficacy study. J Prev Interv Community. 2011;39(2):149-66. doi: 10.1080/10852352.2011.556573. PMID 21480032